CLINICAL TRIAL: NCT04470219
Title: Digital Support for People With Cognitive Impairment - an Intervention to Increase Occupational Performance and the Possibility to Live a More Independent Life
Brief Title: Digital Support for People With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Tiny Jaarsma, Professor at the Faculty of Medicine and Health Sciences, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RemindMe
Record Dates: First submitted 2020-03-27; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Cognitive Impairments; Stroke; Brain Injuries
Keywords: Self-Help Devices; Occupational Therapy
MeSH Terms: conditions — Cognitive Dysfunction; Stroke; Brain Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants receive rehabilitation as usual and training how to use RemindMe by personnel from the research group and an occupational therapist working at the rehabilitation clinic. The participants will use RemindMe for two months. The participants choose activities that he/she wishes to remember to carry out with support by RemindMe. An individual follow-up session will be conducted once a week by the occupational therapist to evaluate if the chosen activities were performed and discuss strategies for the continued use of RemindMe. After two months the participants decide if he/she wants to continue to use RemindMe.
  Interventions: Other: Cognitive support by RemindMe
- control group (No Intervention): The control group receive treatment as usual by the rehabilitation personnel, for example, occupational therapists give interventions that provide support for memory, it could be a paper calendar or other memory devices or strategies.

INTERVENTIONS:
Other: Cognitive support by RemindMe
  Arms: intervention group

SUMMARY:
Cognitive impairment may cause problems in planning and initiating daily activities, as well as remembering to do what is scheduled. This study investigates the effectiveness of an interactive web-based mobile reminder calendar, (RemindMe). The calendar sends text messages to the user's mobile phone as support in everyday life, for persons with cognitive impairment due to neurological injury/diagnoses. The study has a randomized controlled trial design with data collection at baseline and at follow-up sessions after two and four months. Data collection started in October 2016 and continued until February 2018. RemindMe may give the needed support to remind the person and thus increase the ability to perform activities and to become independent in everyday life.

ELIGIBILITY:
Inclusion Criteria:

* Participants with cognitive impairment after stroke or other neurological diseases/injury
* Participants experiencing the need for support in planning, organizing and remembering to do activities in everyday life
* Participants having access to a computer and mobile phone/smartphone
* Participants having linguistic ability to participate in assessments

Exclusion Criteria:

* Participants with palliative care needs
* Participants with reduced vision and/or hearing loss that affects the ability to use a mobile phone/smartphone
* Participants with depression or psychiatric illness

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Occupational performance is assessed at baseline. Change from baseline in occupational performance is assessed after two months. And change from baseline after four months.
  The assessment is used to identify and measure performance and satisfaction with the performance of activities of daily living that are important to the person. Assessment is made on a scale from 1 to 10. 1 is the worst outcome and 10 is the best outcome.
Functional independence measure (FIM) | Independence is assessed at baseline. Change from baseline in independence is assessed after two months. And change from baseline after four months.
  The assessment is used to identify and measure independence in everyday Life activities. Assessment is made on a scale from 1 to 7. 1 is the worst outcome and 7 is the best outcome.

SECONDARY OUTCOMES:
EQ-5D-5L | HQoL is assessed at baseline. Change from baseline in HQoL is assessed after two months. And change from baseline after four months
  The assessment is used to assess Health-related Quality of Life (HQoL). Assessment is made on a Visual Analog Scale from 1 to 100. 1 is the worst outcome and 100 is the best outcome.
Psychosocial Impact of Assistive Device Scale (PIADS) | The psychosocial impact is assessed at baseline. Change from baseline in psychosocial impact is assessed after two months. And change from baseline after four months.
  The assessment is used to assess an Assistive Device Psychosocial impact on a person. Assessment is made on a scale from -3 to 3. -3 is the worst outcome, 0 is neutral impact and 3 is the best outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tiny Jaarsma, Principal Investigator — Faculty of Medicine and Health Sciences Linkoping University
Locations (1):
- Region of Ostergotland, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Study result will be presented in Peer reviewed Open access journal